CLINICAL TRIAL: NCT06462729
Title: A Randomized Study of LDGraft in Single Level Anterior Lumbar Interbody Fusion (ALIF)
Brief Title: LDGraft in Single Level Anterior Lumbar Interbody Fusion (ALIF)
Acronym: RESTORE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Locate Bio Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Locate Bio Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI-001
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease; Lumbar Disc Disease; Spine Disease; Lumbar Spine Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral disc disease; Spinal Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, single-blind, dose-finding, multi-center study which intends to demonstrate the safety of both LDGraft groups versus allograft during a single level ALIF procedure.
  The study will enrol patients with lumbar degenerative disc disease (DDD) requiring single level ALIF. After a screening period, qualified participants will be enrolled and randomized using a 3:3:2 ratio to receive the LDGraft or the control treatment-allograft bone via spinal surgery and will then complete the safety follow-up period.
Who Masked: Participant
Masking Description: Participants will be blinded to the treatment assigned and received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- LDGraft 0.5mg/cc (Experimental)
  Interventions: Device: LDGraft
- LDGraft 1.0mg/cc (Experimental)
  Interventions: Device: LDGraft
- Control Allograft Bone (Active Comparator)
  Interventions: Other: Allograft Bone

INTERVENTIONS:
Device: LDGraft — LDGraft 0.5mg/cc rhBMP-2 applied within intervertebral cage with placement of anterior fixation (plate and screws)
  Arms: LDGraft 0.5mg/cc
Device: LDGraft — LDGraft 1.0mg/cc rhBMP-2 applied within intervertebral cage with placement of anterior fixation (plate and screws)
  Arms: LDGraft 1.0mg/cc
Other: Allograft Bone — Allograft bone (100% human tissue product) applied within intervertebral cage with placement of anterior fixation (plate and screws)
  Arms: Control Allograft Bone

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of LDGraft (investigational device) compared to 100% human tissue product allograft bone (control) when applied in an ALIF procedure in the treatment of patients with lumbar degenerative disc disease (DDD).

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, single-blind, dose-finding, multi-center study which intends to demonstrate the safety of both LDGraft groups versus allograft during a single level ALIF procedure. This is a first in human (FIH) study.

The study will enroll patients with lumbar degenerative disc disease (DDD) requiring single level ALIF. The procedure will involve use of an intervertebral cage and fixation (plate and screws).

Upon successful completion of the Screening period and confirmation of eligibility the participant will allocated 3:3:2 to the LDGraft groups (investigational) or the allograft control group. Participants will be blinded to the treatment assigned however the surgical procedure and the post operative recovery will be managed in accordance with standard clinical practice for anterior lumbar interbody fusion.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature adults ≥22 and ≤80 years at the time of surgery
2. Willing and able to give written informed consent and comply with study protocol and postoperative management program
3. Degenerative disc disease of the lumbosacral spine in one level (L3 to S1) requiring fusion confirmed by patient history and radiographic imaging (CT/MRI/X-rays) with one or more of the following:

   * instability (as defined by ≥3mm translation or ≥5° angulation);
   * osteophyte formation of facet joints or vertebral endplates;
   * decreased disc height, on average by >2mm, but dependent upon the spinal level;
   * scarring/thickening of ligamentum flavum, annulus fibrosis, or facet joint capsule;
   * herniated nucleus pulposus;
   * facet joint degeneration/changes; and/or
   * vacuum phenomenon.
4. Preoperative Oswestry Disability Index score ≥ 35
5. Participant has not responded to conservative treatment (e.g. medications, injections, physical therapy, etc.) for a period of 6 months
6. Participant is indicated for an ALIF approach to the lumbar spine

Exclusion Criteria:

1. Previous lumbar spine instrumentation (i.e., anterior disc replacement, interspinous device) or a previous interbody fusion procedure in the lumbar spine
2. More than one level lumbar spine level requiring fusion
3. Three or more contiguous lumbar spine levels requiring decompression (Note: Up to two contiguous levels of decompression is acceptable)
4. Known hypersensitivity or allergy to any components of the study treatments inclusive of hypersensitivity or allergy to any BMP-2 type recombinant proteins or peptides.
5. Pregnant, planning to become pregnant during the follow-up time period, or breast-feeding women
6. Presence of active malignancy
7. Requires bone growth stimulation in the lumbar spine
8. Active local or systemic infection
9. Spondylolisthesis greater than Grade 1 (25% translation)
10. Currently smoking or using nicotine products, including e-cigarette products (e.g., vaping) (Use within 30 days of screening date is considered 'current')
11. Any degenerative muscular or neurological condition that would interfere with evaluation of outcomes, including but not limited to Parkinson's disease, amyotrophic lateral sclerosis (ALS), or multiple sclerosis
12. Any medical condition requiring treatment with any drug known to potentially interfere with bone/soft tissue healing (e.g. chronic systemic steroids) or receiving radiation therapy that is expected to continue for the duration of the study
13. Body Mass Index > 35
14. Insulin-dependent diabetes mellitus
15. Osteopenia or osteoporosis of the spine, DEXA T score of ≤ -1.0
16. Any secondary causes of osteoporosis (e.g. chronic liver or kidney disease, uncontrolled hyper- or hypothyroidism, type I or type II diabetes mellitus, gastrointestinal malabsorption syndromes) or other conditions known to adversely affect osteogenesis (e.g. Paget's disease, Ehlers-Danlos syndrome or osteogenesis imperfecta)
17. Participation in another investigational study within 30 days prior to surgery for investigational devices, or within the last three months for investigational drugs;
18. Current or recent history of chemical/alcohol abuse or dependency using standard medical definition of DSM-5 (Diagnostic and Statistical Manual) code
19. In the opinion of the investigator, the participant has a behavioral, cognitive, social or medical problem that may interfere with the assessment of the safety or effectiveness of the product
20. Radiographically compromised vertebral bodies at the index level due to current or past trauma, e.g., by the radiographic appearance of the fracture callus, deformity, malunion or nonunion
21. Currently a prisoner
22. Involved in active litigation relating to his/her spinal condition or workers compensation claimants.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion | 12 months and 24 months
  Radiographic fusion defined as evidence of bridging bone by CT scan
Secondary Surgical Intervention | 12 months and 24 months
  No index level secondary surgical intervention
Oswestry Disability Index (ODI) Score | 12 months and 24 months
  At least 15-point improvement in Oswestry Disability Index (ODI) compared to baseline
Neurological Condition | 12 months and 24 months
  No new or worsening persistent lumbar spine neurological condition compared to baseline
Serious Device-Related Adverse Events | 12 months and 24 months
  No serious device-related adverse events

SECONDARY OUTCOMES:
Radiographic Outcomes | 6 weeks, 3 months, 6 months, 12 months and 24 months
  Radiographic outcomes including bridging bone, radiolucency, device condition, migration, subsidence, angular motion, and translational motion
Visual Analog Score (VAS) Back | 6 weeks, 3 months, 6 months, 12 months and 24 months
  Improvement in the Visual Analog Score (VAS) back pain of 20mm compared to baseline
Visual Analog Score (VAS) Change Back | 6 weeks, 3 months, 6 months, 12 months and 24 months
  Mean change in back VAS over time intervals
Visual Analog Score (VAS) Leg | 6 weeks, 3 months, 6 months, 12 months and 24 months
  Improvement in the Visual Analog Score (VAS) worst leg of 20mm compared to baseline
Visual Analog Score (VAS) Change Leg | 6 weeks, 3 months, 6 months, 12 months and 24 months
  Mean change in leg VAS over time intervals
Oswestry Disability Index (ODI) Score | 6 weeks, 3 months, 6 months, 12 months and 24 months
  Improvement in ODI of 15 points compared to baseline
Oswestry Disability Index (ODI) Change | 6 weeks, 3 months, 6 months, 12 months and 24 months
  Mean change in ODI over time intervals

CONTACTS AND LOCATIONS:
Locations (3):
- Orthopaedics NorthEast, Fort Wayne, Indiana, United States
- Australia (2):
  - Newcastle Private Hospital, Newcastle, New South Wales
  - Macquarie University, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No